CLINICAL TRIAL: NCT05003362
Title: Acceptance and Commitment Therapy for High Frequency Episodic Migraine
Brief Title: ACT for High Frequency Migraine; A Virtual Mindfulness Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Massachusetts Institute of Technology (Other)
Responsible Party: Principal Investigator, Carolyn A. Bernstein, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2018P001239
Record Dates: First submitted 2021-07-20; First posted 2021-08-12 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Migraine
Keywords: migraine; high frequency; ACT
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Intervention Model Description: After screening, patients will be randomized and one group will receive the intervention. The investigators will do sequential interventions of the ACT
Who Masked: Outcomes Assessor
Masking Description: randomized control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- usual care (No Intervention): Subjects randomized to the usual care control group will continue using their usual medical care as prescribed by their physician.
- ACT (Active Comparator): An 8-week mindfulness-based group therapy.
  Interventions: Behavioral: ACT

INTERVENTIONS:
Behavioral: ACT — mindfulness intervention for patients with pain/migraine
  Arms: ACT

SUMMARY:
Mindfulness Training specifically for pain to be offered to migraine patients

DETAILED DESCRIPTION:
Patients with high frequency migraine will be randomized to UC or intervention. Those in intervention will attend a multi session training on Acceptance and Commitment Therapy. All participants will track responses.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 18-65
* Diagnosis of episodic migraine (according to International Classification for Headache Diagnosis criteria)
* 4-14 migraine days per month over the past 3 months
* No change in medication in the past 3 months
* Greater than 1 year of migraines
* Agreeable to participate, commit to all study procedures and to be randomized to either group
* Fluent in English

Exclusion Criteria:

* Any unstable medical or psychiatric conditions requiring immediate treatment or could lead to difficulty complying with the protocol
* Active suicidal ideation
* Moderate to severe depression
* Current alcohol or substance abuse
* Recent Cognitive Behavioral Therapy, Mindfulness Based Cognitive Therapy, Dialectic Behavioral Therapy or Acceptance and Commitment Therapy within past 3 years
* Current use of narcotics
* Psychiatric hospitalization within past year
* Comorbid pain condition rated as more painful than migraine
* Starts new migraine treatment during study
* Inability to complete study visits

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — patients will identify as female
Enrollment: 75 (Actual)
Dates: Start 2020-10-25 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2021-11-23 (Actual)

PRIMARY OUTCOMES:
Feasibility of a randomized controlled trial of ACT | one year
  Demonstrate that 48 patients can be successfully enrolled and randomized

SECONDARY OUTCOMES:
Preliminary data on the effectiveness of ACT on migraine frequency and migraine disability | one year
  Patient-completed migraine logs will be used to record the number of migraine days/month. Migraine disability will be measured using the validated Migraine Disability Assessment (MIDAS) questionnaire.
Change in migraine severity, duration, and medication use. | one year
  Severity of each migraine (1-10), duration (hours), and medicines taken assessed by patient-completed migraine logs.
Change in headache-related disability | one year
  Headache Related Disability measured using the validated HIT-6.
Change in quality of life. | one year
  Quality of life assessed using the Migraine Specific Quality of Life Questionnaire (MSQ).
Change in depression and anxiety. | one year
  Depression and anxiety assessed through the Hospital Anxiety and Depression Scale (HADS).
Change in pain acceptance and pain expectancy. | one year
  Pain acceptance assessed through the Chronic Pain Acceptance Questionnaire and pain expectancy during the migraine attacks assessed using the allodynia questionnaire.
Change in pain catastrophizing. | one year
  Pain Catastrophizing Scale (PCS) used to assess distress and rumination experienced due to migraine anticipation.
Change in distress tolerance. | one year
  Distress tolerance will be assessed through the Distress Tolerance Scale.
Change in physical activity. | one year
  Physical activity measured using the Godin Leisure Time Exercise questionnaire.
Change in perceived stress. | one year
  Perceived stress measured through the Perceived Stress Scale (PSS).
Change in mindfulness. | one year
  Mindful Attention and Awareness Scale (MAAS) used to measure receptive awareness and attention to the present.
Change in cortisol levels. | one year
  Salivary Cortisol will be collected to measure the cortisol awakening response.

CONTACTS AND LOCATIONS:
Overall Officials: carolyn bernstein, md, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Womens Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bernstein C, Lazaridou A, Paschali M, Vilsmark ES, Rist PM. Acceptance-Commitment Therapy for Women with Episodic Migraine: A Pilot Randomized Trial. J Integr Complement Med. 2024 May;30(5):478-486. doi: 10.1089/jicm.2023.0085. Epub 2023 Nov 27. PMID 38011750